CLINICAL TRIAL: NCT03613090
Title: Novel Collagen Scaffold vs Conventional Scaffold in Regeneration of Human Dental Pulp Tissue
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn-was not approved by IRB
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Collagen Matrix (Industry)
Responsible Party: Principal Investigator, David Clanton DMD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-161031003
Record Dates: First submitted 2018-06-19; First posted 2018-08-02 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Root Canal Therapy

STUDY DESIGN:
Intervention Model Description: Investigators will screen routine root canal treatment-seeking patients who present normally to clinic as potential study participants. The patients selected will be those who will require root canal therapy as a part of their routine dental care.
  Participant will be randomly assigned to one or two groups:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Collagen-hydroxyapatite Scaffold (Syn-Oss) (Experimental): Placement of a collagen-hydroxyapatite scaffold (Syn-Oss), placement of a tricalcium silicate barrier (mineral trioxide aggregate), placement of a composite occlusal restoration (standard dental material).
  Interventions: Drug: Collagen-hydroxyapatite scaffold (Syn-Oss)
- Collagen Scaffold (Colla-Plug) (Active Comparator): Placement of a collagen scaffold (Colla-Plug) over a blood clot, placement of a tricalcium silicate barrier (mineral trioxide aggregate), placement of a composite occlusal restoration (standard dental material). The Colla-Plug material is placed adjacent to the blood clot that has formed inside the root canal space. It act as a matrix for the subsequent placement of the mineral trioxide aggregate material. It has been used as the standard of care in regenerative endodontics since 2004.
  Interventions: Drug: Collagen Scaffold (Colla-Plug)

INTERVENTIONS:
Drug: Collagen-hydroxyapatite scaffold (Syn-Oss) — The aim of this study is to add to the existing body of regenerative endodontics research by providing human radiographic evidence for the healing process which occurs after the placement of a FDA-approved collagen-hydroxyapatite scaffold, in the use of a blood clot
  Arms: Collagen-hydroxyapatite Scaffold (Syn-Oss)
Drug: Collagen Scaffold (Colla-Plug) — Traditionally, endodontic therapy consisted of removing the infected dental pulp from the canal spaces and replacing it with an artificial substitute called gutta percha. Regenerative endodontic research efforts were originally concentrated upon treatment of the immature necrotic tooth whereby stem cells from the bone near the root end were stimulated to grow onto a blood clot scaffold created within the debrided and disinfected canal space. The hope is that the stem cells would differentiate into cells which could potentially replace the lost pulpal tissues, restoring what was lost due to infection.
  Arms: Collagen Scaffold (Colla-Plug)

SUMMARY:
The purpose of this investigation is to assess the use of a novel scaffold (an FDA-approved collagen-hydroxyapatite material called Syn-Oss) for regeneration of pulp tissues versus the use of a traditional scaffold (blood clot).

DETAILED DESCRIPTION:
Regeneration of pulp tissues in teeth with immature roots is a new concept based on historical limited success using calcium hydroxide dressings placed into debrided pulp spaces. Obtaining stem cells from the apical papilla (SCAP cells), which are present at the base of all teeth, but are most accessible in teeth with immature apices, greatly enhances clinical success. Current therapies lack ideal messenger chemicals and scaffolds to optimize results.

ELIGIBILITY:
Inclusion Criteria:

1. Single root canal space apparent on a standard dental periapical radiograph
2. Immature tooth apex width at least 1.1mm in diameter as measured from the radiograph
3. No history of antibiotic drug allergy
4. Necrotic pulp as demonstrated by coronal discoloration.
5. Periapical radiolucency
6. Negative pulp sensibility tests
7. Other standard clinical means of assessing pulp vitality status

Exclusion Criteria:

1. Any patients having an American Association of Anesthesiologists 4 health classification will be excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Observation 1-Radiodensity at apex @ 1mm from root vertex | Month 0-3, Institutional Review Board proposal and approval
  Grade 1 = no disruption of apical anatomy Grade 2 = Periodontal ligament (PDL) width double thickness, with intact lamina dura Grade 3 = break in lamina dura
Observation 2 - Increase in dentin wall thickness. It is noted that minimal change is expected over the course of this short-term study. | Months 3-6, patient recruitment and revascularization surgery in Department of Endodontics
  Grade 1 = dentin wall thickness increased by > 1mm Grade 2 = dentin wall thickness < 1mm
Observation 3 - Increase in root length, in mm. | Month 6-12, clinical and radiographic recall and assessment
  Grade 1 = root length increased > 1 mm Grade 2 = root length increased 0-1 mm Grade 3 = root length shorter than pre-op
Observation 4 - Periradicular status | Month 13-15, data analysis and manuscript preparation
  Grade 1 = no periradicular radiolucency Grade 2 = periradicular radiolucency 0-1 mm in diameter Grade 3 = periradicular radiolucency > 1 mm in diameter

CONTACTS AND LOCATIONS:
Overall Officials: David Clanton, DMD, Principal Investigator — Univeristy of Alabama at Birmingham; Paul D Eleazer, DDS, Principal Investigator — Univeristy of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States